CLINICAL TRIAL: NCT02117193
Title: Combined and Isolated Effects of Sleep Deprivation and Alcohol Intake on Cardiorrespiratory, Neuromuscular and Hormonal Responses in Healthy Males.
Brief Title: Combined and Isolated Effects of Sleep Deprivation and Alcohol Intake on Exercise Performance in Humans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Marco Aurélio Vaz, PhD, PhD, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: UFRGS 366465
Record Dates: First submitted 2014-04-14; First posted 2014-04-17 (Estimated); Results first posted 2016-09-22 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-10

CONDITIONS: Alcohol Intake; Sleep Deprivation
MeSH Terms: conditions — Alcohol Drinking; Sleep Deprivation | interventions — Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alcohol intake (Placebo Comparator): 1 g/kg of etanol combined. Beer without alcohol in the same volume will be used to placebo condition.
  Interventions: Other: Alcohol intake; Other: Sleep deprivation
- sleep deprivation (Active Comparator): one night of sleep deprivation will be compared to 8h of normal sleep.
  Interventions: Other: Alcohol intake; Other: Sleep deprivation

INTERVENTIONS:
Other: Alcohol intake — The subjects will be drink beer (with or without alcohol) before sleep intervention (normal sleep and sleep deprivation).
Other: Sleep deprivation — One night of sleep deprivation or one night of normal sleep.

SUMMARY:
Although the effects of acute alcohol intake and sleep deprivation on exercise performance lacks evidence in the literature, in many situations, they occur simultaneously. Once the alcohol affects physiological processes, the processes that occur during sleep can be impaired, such as: suppression of GH release, action of neurotransmitters and neuromodulators in the CNS, changes in the proportion of sleep stages and may lead to suppression of REM sleep. These changes promote a significant functional impairment such as a reduction in alertness and modification in reaction time, which affects the performance of any activity of daily and professional life. However, the combined effects on the physical performance variables, such as aerobic and neuromuscular performance lack of evidence in the literature.

DETAILED DESCRIPTION:
Ten subjects were randomized in four situations after familiarization and control situation: (1) alcohol intake combined with sleep normal; (2) alcohol intake combined with sleep deprivation; (3) placebo intake combined with sleep normal and (4) placebo intake combined with sleep deprivation.

ELIGIBILITY:
Inclusion Criteria:

- Physical active men

Exclusion Criteria:

* AUDIT questionnaire above 15 points
* Nocturnal Chronotype
* Skeletal muscle injuries in upper and lower limb
* Metabolic and cardiovascular disease

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Rodrigues, MSc, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Exercise Research Laboratory, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: This is a cross-over study.
Period: Overall Study
Arm/Group | All Study Participants
Started | 10
Alcohol Intake + Normal Sleep | 10
Placebo Intake + Normal Sleep | 10
Alcohol Intake + Sleep Deprivation | 10
Placebo Intake + Sleep Deprivation | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Received Alcohol intake + Normal Sleep Received Alcohol intake + Sleep Deprivation Received Placebo intake + Normal Sleep Received Placebo intake + Sleep Deprivation
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.5 (3.3)
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  Brazil | 10
maximal oxygen uptake [Mean (Standard Deviation); unit: ml.kg-1.min-1] | 44.8 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Aerobic Performance
Description: Aerobic performance will be determined through the subject's heart rate
Time Frame: After each sequence, up to 8 hours
Measure: Mean (Standard Deviation); unit: bpm
Groups:
- Sequence 1: Alcohol intake + Normal Sleep
  Alcohol intake: The subjects will be drink beer (1g/kg of ethanol) before sleep.
  Normal sleep: One night of normal sleep (8h)
- Sequence 2: Alcohol intake + Sleep deprivation
  Alcohol intake: The subjects will be drink beer (1g/kg of ethanol) before sleep.
  Sleep deprivation: One night of sleep deprivation (8h)
- Sequence 3: Placebo intake + Normal Sleep
  Placebo intake: The subjects will be drink beer (zero alcohol) before sleep.
  Normal sleep: One night of normal sleep (8h)
- Sequence 4: Placebo intake + Sleep deprivation
  Placebo intake: The subjects will be drink beer (zero alcohol) before sleep.
  Sleep deprivation: One night of sleep deprivation (8h)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Number analyzed (Participants) | 10 | 10 | 10 | 10
bpm | 172 (12.19) | 173 (9.2) | 175 (6.5) | 176 (11.4)

2. Primary Outcome: Neuromuscular Performance
Description: knee extensor isometric torque
Time Frame: After each sequence, up to 8 hours
Measure: Mean (Standard Deviation); unit: Nm
Groups:
- Sequence 1: Alcohol intake + Normal Sleep
  Alcohol intake: The subjects will be drink beer (1g/kg ethanol) before sleep.
  Normal sleep: One night of normal sleep (8h)
- Sequence 2: Alcohol intake + Sleep deprivation
  Alcohol intake: The subjects will be drink beer (1g/kg ethanol) before sleep.
  Sleep deprivation: One night of sleep deprivation (8h)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Number analyzed (Participants) | 10 | 10 | 10 | 10
Nm | 260.8 (27.9) | 242.3 (34.3) | 258.9 (31.3) | 249.5 (33.9)

3. Primary Outcome: Biochemical Responses
Description: Glucose after each situation in the morning
Time Frame: After each sequence, up to 8 hours
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Alcohol Intake + Normal Sleep: 1g/kg of alcohol (beer) combined with 8 hours of normal sleep
- Alcohol Intake + Sleep Deprivation: 1g/kg of alcohol (beer) combined with 8 hours of sleep deprivation
- Placebo Intake + Normal Sleep: Placebo (beer without alcohol in the same volume to beer with alcohol) combined with 8 hours of normal sleep
- Placebo Intake + Sleep Deprivation: Placebo (beer without alcohol in the same volume to beer with alcohol) combined with 8 hours of sleep deprivation
Arm/Group | Alcohol Intake + Normal Sleep | Alcohol Intake + Sleep Deprivation | Placebo Intake + Normal Sleep | Placebo Intake + Sleep Deprivation
Number analyzed (Participants) | 10 | 10 | 10 | 10
mg/dl | 89.82 (6.60) | 84.76 (4.03) | 92.77 (5.13) | 92.85 (8.26)

4. Secondary Outcome: Hydration Status
Description: Urine Specific Gravity
Time Frame: After each sequence, up to 8 hours
Measure: Mean (Standard Deviation); unit: g/ml
Groups:
- Sequence 3: Placebo intake + Normal Sleep
  Placebo intake: The subjects will be drink beer (zero alcohol, in the same volume that alcohol intake) before sleep.
  Normal sleep: One night of normal sleep (8h)
- Sequence 4: Placebo intake + Sleep deprivation
  Placebo intake: The subjects will be drink beer (zero alcohol, in the same volume that alcohol intake) before sleep.
  Sleep deprivation: One night of sleep deprivation (8h)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Number analyzed (Participants) | 10 | 10 | 10 | 10
g/ml | 1.017 (0.006) | 1.017 (0.005) | 1.015 (0.003) | 1.011 (0.006)

5. Secondary Outcome: Profile of Mood States
Time Frame: 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Breath Alcohol
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Alcohol Intake + Normal Sleep: 1 g/kg of etanol combined with 8 hours of normal sleep
- Alcohol Intake + Sleep Deprivation: 1 g/kg of etanol combined with 8 hours of sleep deprivation
Arm/Group | Alcohol Intake + Normal Sleep | Alcohol Intake + Sleep Deprivation | Placebo Intake + Normal Sleep | Placebo Intake + Sleep Deprivation
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 8/10 | 0/10 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alcohol Intake + Normal Sleep (N=10) | Alcohol Intake + Sleep Deprivation (N=10) | Placebo Intake + Normal Sleep (N=10) | Placebo Intake + Sleep Deprivation (N=10)
Fatigue (Nervous system disorders) | 5 | 8 | 0 | 3
Headache (Nervous system disorders) | 5 | 8 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes